CLINICAL TRIAL: NCT04682951
Title: Good Prognosis Factors After Decompressive Craniectomy : a Ten-year Retrospective Study
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, AUDIBERT Gérard, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2020PI244
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Decompressive Craniectomy; Brain Injuries; Treatment Outcome
Keywords: Decompressive craniectomy; Outcome; Brain injuries; Aneurysmal subarachnoid hemorrhage; Cerebral venous thrombosis; Intracerebral hemorrhage; Ischemic stroke; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries; Subarachnoid Hemorrhage; Intracranial Thrombosis; Cerebral Hemorrhage; Ischemic Stroke; Brain Injuries, Traumatic | interventions — Decompressive Craniectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Decompressive Craniectomy

SUMMARY:
Decompressive craniectomy is a treatment of refractory intracranial hypertension after various etiologies : malignant ischemic stroke, traumatic brain injury, intraparenchymal hemorrhage, aneurysmal subarachnoid hemorrhage, cerebral venous thrombosis.

Initially considered as a lifesaving therapy, benefits in terms of survival were shown compared to medical treatment alone.

However, despite a better survival, morbidity and poor neurological outcome are frequent among survivors.

The objective of the study is to identify initial good neurological outcome factors after decompressive craniectomy in a large series of patients, in order to argue surgical and intensive care decisions, considering expected benefit and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a decompressive craniectomy from 06/11/2008 to 06/15/2018 in CHRU Nancy, France.

Exclusion Criteria:

* Infectious ou malignant disease leading to decompressive craniectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a decompressive craniectomy on a 10 year period in CHRU Nancy, France.
Sampling Method: Non-Probability Sample
Enrollment: 544 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Good neurological outcome | 6 months after surgery
  The neurological outcome is considered "good" when Glasgow Outcome Score extended (GOSE) assessed 6 months after decompressive craniectomy is between 5 and 8.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No